CLINICAL TRIAL: NCT05810649
Title: Local Injection Freshly Manufactured 35kDa Hyaluronan Fragment HA35 for Treatment of Chronic Wounds and Pain Caused by Chronic.
Brief Title: Local Injection for the Treatment of Chronic Wounds and Pain Caused by Chronic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nakhia Impex LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSHN002
Record Dates: First submitted 2023-03-31; First posted 2023-04-12 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-03

CONDITIONS: Pain; Chronic Wound
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HA35 local injection Group (Experimental): This clinical study used the 35 kDa low molecular weight HA fragment HA35, which was freshly manufactured by mixing bovine testis-derived hyaluronidase PH20 injection (H31022111) with high-molecular-weight HA injection (H20174089) for 20 minutes at room temperature.
  Interventions: Drug: Freshly manufactured 35 kDa hyaluronan fragment

INTERVENTIONS:
Drug: Freshly manufactured 35 kDa hyaluronan fragment — One hundred milligrams of the freshly made 35 kDa low molecular weight HA fragment HA35 was injected into the tissue under the heath skin immediately surrounding the chronic wounds once a day for 10 days.The pain associated with the wounds and degree of wound healing, including the size of the fresh granulation area on the wound; the degree to which the surface of the skin surrounding the wound was dark, red, dry or broken; and the size of the wound, were observed and recorded.
  Other Names: HA35

SUMMARY:
Chronic wounds are wounds or ulcers that do not heal properly and are generally classified as venous, arterial, diabetic, traumatic and pressure chronic wounds and is often associated with inflammatory and neuropathic pain. Preliminary clinical studies have confirmed that injection of freshly prepared HA35 promoted the healing of chronic wounds and relieved the pain associated with chronic wounds. This clinical study is a prospective repeated experiments. The purpose of this study was to verify the effectiveness of HA35 injection therapy.

DETAILED DESCRIPTION:
Our previous study, together with other studies, showed that topical use of the tissue-permeable HA fragment HA35 relieves swelling of the skin and mucosal wounds. In this study, the tissue-permeable 35 kDa HA fragment HA35 was freshly manufactured by mixing hyaluronidase PH20 injectable solution (H31022111) and high-molecular-weight HA injectable solution (H20174089). The therapeutic effect of the tissue-permeable HA fragment HA35 for the treatment of pain-associated chronic wounds was studied in a single-arm off-label study before and after treatment comparison.

ELIGIBILITY:
Inclusion Criteria:

* The chronic wounds of painful diabetic wounds, venous wounds, arterial wounds, traumatic and pressure wounds whichvhad not been closed more than 3 months.
* All the chronic wounds were clinically presented by surface darkeness and purulent secretions on the wounds, and darkness or redness, swelling, dryness and broken surface of the skin immediately surrounding the wounds.
* Subject agrees to be compliant with study related visit and treatment schedule.
* Written informed consent.
* Adults aged 18-60 years.

Exclusion Criteria:

* Have a persistent pain resulted from other medical conditions or unknown causes.
* History of wound healing abnormalities or a medical condition that is known to be associated with abnormal wound healing.
* Subjects with any known coagulation disorder.
* Pregnant females.
* Be concomitantly participating in another clinical study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-02 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
Wound-associated pain measurement | 24 hours
  Each participant rated the pain on a scale of 0-10, where 0 represents "no pain" and 10 represents "the most intense pain".
Measurement of darkness or redness of the skin surrounding the wounds | 10 days
  This participant self-assessment scale was used to compare the darkness or redness of the skin surrounding the wounds before and after treatment. The participant then rated the intensity level using a scale of 0-10, where 0 represents "no" and 10 represents "the most".
Measurement of dryness and broken areas of the surface of the skin surrounding the wounds | 10 days
  This participant self-assessment scale was used to compare the dryness and broken areas of the surface of the skin surrounding the wounds before and after the treatment. The participants then rated the intensity level using a scale of 0-10, where 0 represents "no" and 10 represents "the most".
Measurement of fresh granulation growth on the wounds | 10 days
  This participant self-assessment scale was used to compare the fresh granulation growth on the surface of the wounds before and after treatment. The participants then rated the intensity level using a scale of 0-10, where 0 represents "no" and 10 represents "the most".
Measurement of wound size | 10 days
  This participant self-assessment scale was used to compare the size of the wounds before and after the treatment. The participants then rated the size or area using a scale of 0-10, where 0 represents "no" and 10 represents "the most".

CONTACTS AND LOCATIONS:
Locations (1):
- Huinuode Biotechnology Co., Ltd., Qingdao, China